CLINICAL TRIAL: NCT00119912
Title: Norwegian Colorectal Cancer Prevention Trial
Brief Title: NORCCAP: Norwegian Colorectal Cancer Prevention Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian Department of Health and Social Affairs (Other Government)
Collaborators: Norwegian Cancer Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NORCCAP-1; Shdir 97/08614 (Other: Norwegian Department of Health)
Record Dates: First submitted 2005-07-06; First posted 2005-07-14 (Estimated); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Colorectal Cancer; Adenoma
Keywords: screening; flexible sigmoidoscopy; fecal occult blood; cancer; colon; rectum
MeSH Terms: conditions — Colorectal Neoplasms; Adenoma; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A 1 Intervention arm Flex Sig (Active Comparator): Randomised from the population registry, age 50-64 years and invited for Flexible Sigmoidoscopy (Flex Sig) screening. Half of invitees are additionally invited to provide a stool sample for fecal occult blood testing (Intervention arm A 2). They are drawn directly from the population registry without prior consent to be randomized - approved by Regional Ethics Committees of South-East Norway..
  Interventions: Procedure: A 1 Intervention arm Flex Sig
- B Control arm (No Intervention): "No screening group" randomised from population age 50-64 years. As for the active intervention arm, the control group was not informed about being randomized to 'no screening' since 'no screening' was the current usual care (and still is in 2015) in Norway - approved by Regional Ethics Committees of South-East Norway.
- A 2 Intervention arm Flex Sig + iFOBT (Active Comparator): Randomised from the population registry, age 50-64 years and invited for Flexible Sigmoidoscopy (Flex Sig) screening plus an immunochemical test for fecal occult blood (iFOBT). As for arms A 1 and B, they are drawn directly from the population registry without prior consent to be randomized.
  Interventions: Procedure: A 2 Intervention arm Flex Sig + iFOBT

INTERVENTIONS:
Procedure: A 1 Intervention arm Flex Sig — Screening by flexible sigmoidoscopy
  Arms: A 1 Intervention arm Flex Sig
Procedure: A 2 Intervention arm Flex Sig + iFOBT — In addition to Flexible Sigmoidoscopy, half of arm A (randomised 1:1) is invited to provide stool samples for FOBT
  Arms: A 2 Intervention arm Flex Sig + iFOBT

SUMMARY:
The purpose of this study is to see if screening with flexible sigmoidoscopy (a flexible viewing tube) may reduce large bowel cancer and cancer deaths. The researchers also want to see if the addition of screening for occult blood in stools may contribute further to this aim. Additionally, the researchers also want to see to which extent (and in which direction) the study may influence overall endoscopic activity in the general population in the screening area and in areas where controlled screening is not established.

DETAILED DESCRIPTION:
Although flexible sigmoidoscopy (FS) as a screening tool has a much higher test sensitivity than fecal occult blood tests (FOBT) for colorectal cancer and high-risk adenomas, randomised trials with long-term follow-up are missing. The primary aim is to evaluate the effect on CRC mortality and morbidity by screen detection of CRC and removal of precursor lesions (polypectomy of adenomatous polyps)

Secondary aims:

1. Evaluation of cost/effectiveness of screening for CRC and significant, benign lesions using flex-sig only compared to flex-sig in combination with faecal tests
2. To evaluate to which extent (and in which direction) the study may influence overall endoscopic activity in the general population in the screening areas and in areas where controlled screening is not established
3. Determine the prevalence of known types familial CRC in a general population and try to define other groups with intermediate increased risk
4. Clarify possible psychosocial effects of endoscopic screening and how it may influence lifestyle and lifestyle related morbidity and overall mortality

Population:

21,000 men and women, aged 50-64 years, living in the city of Oslo or the county of Telemark are drawn by randomisation (approx. 1:5) from the population registry and invited to have a flexible sigmoidoscopy examination. The control group constitutes 79,000 individuals. Those invited for flexible sigmoidoscopy are further randomised (1:1) to bring or not to bring 3 successive stool samples for FOBT on attendance for FS.

Method:

This is a once-only screening concept with bowel cleansing being limited to a 240 ml Sorbitol enema given on attendance. The threshold for work-up colonoscopy is low as a positive screening test is defined as any polyp >9mm, any histologically verified adenoma irrespective of size and a positive FOBT. The screening phase is limited to the period January 1999- January 2002 and the first follow-up results will not be reported until all entries have passed the 5-year mark (i.e. in early 2007).

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* Living in Oslo or Telemark
* Age 50-64 years

Exclusion Criteria:

* Patients with previous open colorectal surgery (resections, enterostomies)
* Individuals in need of long lasting attention and nursing services (somatic or psychosocial reasons, mental retardation)
* On-going cytotoxic treatment or radiotherapy for malignant disease
* Severe chronic cardiac or lung disease (NYHA III-IV)
* Patients with heart valve replacement on life long anticoagulant therapy
* A coronary event during the last 3 months if having lead to hospitalisation
* Cerebrovascular accident during the last 3 months
* Resident abroad

Ages: 50 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100000 (Actual)
Dates: Start 1999-01; Primary Completion 2036-12 (Estimated); Study Completion 2036-12 (Estimated)

PRIMARY OUTCOMES:
1. Evaluate the effect on CRC mortality and morbidity by screen detection of CRC and removal of precursor lesions (polypectomy of adenomatous polyps).First evaluation after 5 years. | Evaluations in 2007 (published),2012,2017
  CRC incidence and mortality is followed

SECONDARY OUTCOMES:
1. Determine the prevalence of known types familial CRC in a general population and try to define other groups with intermediate increased risk. Results "in press" 2005. | Evaluated in 2005 (published)
  Determine the prevalence of familial CRC in a general population sample
2. Clarify possible psychosocial effects of endoscopic screening and how it may influence lifestyle and lifestyle related morbidity and overall mortality. Evaluation in 2005. | Evaluated in 2005 (published)
  Determine psychosocial effects of invitation to screening and of screening findings

CONTACTS AND LOCATIONS:
Overall Officials: Giske Ursin, M.D., Study Chair — Institute of Population-based Cancer Research
Locations (1):
- Institute of Population-based Cancer Research, Oslo, Norway

REFERENCES:
- [Background] Hoff G, Grotmol T, Skovlund E, Bretthauer M; Norwegian Colorectal Cancer Prevention Study Group. Risk of colorectal cancer seven years after flexible sigmoidoscopy screening: randomised controlled trial. BMJ. 2009 May 29;338:b1846. doi: 10.1136/bmj.b1846. PMID 19483252
- [Background] Holme O, Bretthauer M, Eide TJ, Loberg EM, Grzyb K, Loberg M, Kalager M, Adami HO, Kjellevold O, Hoff G. Long-term risk of colorectal cancer in individuals with serrated polyps. Gut. 2015 Jun;64(6):929-36. doi: 10.1136/gutjnl-2014-307793. Epub 2014 Nov 16. PMID 25399542
- [Background] Berstad P, Loberg M, Larsen IK, Kalager M, Holme O, Botteri E, Bretthauer M, Hoff G. Long-term lifestyle changes after colorectal cancer screening: randomised controlled trial. Gut. 2015 Aug;64(8):1268-76. doi: 10.1136/gutjnl-2014-307376. Epub 2014 Sep 2. PMID 25183203
- [Background] Holme O, Loberg M, Kalager M, Bretthauer M, Hernan MA, Aas E, Eide TJ, Skovlund E, Schneede J, Tveit KM, Hoff G. Effect of flexible sigmoidoscopy screening on colorectal cancer incidence and mortality: a randomized clinical trial. JAMA. 2014 Aug 13;312(6):606-15. doi: 10.1001/jama.2014.8266. PMID 25117129
- [Result] Larsen IK, Grotmol T, Almendingen K, Hoff G. Impact of colorectal cancer screening on future lifestyle choices: a three-year randomized controlled trial. Clin Gastroenterol Hepatol. 2007 Apr;5(4):477-83. doi: 10.1016/j.cgh.2006.12.011. Epub 2007 Mar 23. PMID 17363335
- [Result] Larsen IK, Grotmol T, Almendingen K, Hoff G. Lifestyle as a predictor for colonic neoplasia in asymptomatic individuals. BMC Gastroenterol. 2006 Jan 13;6:5. doi: 10.1186/1471-230X-6-5. PMID 16412216
- [Result] Larsen IK, Grotmol T, Almendingen K, Hoff G. Lifestyle characteristics among participants in a Norwegian colorectal cancer screening trial. Eur J Cancer Prev. 2006 Feb;15(1):10-9. doi: 10.1097/01.cej.0000186636.27496.bb. PMID 16374224
- [Result] Stormorken AT, Hoff G, Norstein J, Bowitz-Lothe IM, Hanslien E, Grindedal E, Moller P. Estimated prevalence of hereditary cancers and the need for surveillance in a Norwegian county, Telemark. Scand J Gastroenterol. 2006 Jan;41(1):71-9. doi: 10.1080/00365520510023891. PMID 16373279
- [Result] Gondal G, Grotmol T, Hofstad B, Bretthauer M, Eide TJ, Hoff G. Biopsy of colorectal polyps is not adequate for grading of neoplasia. Endoscopy. 2005 Dec;37(12):1193-7. doi: 10.1055/s-2005-921031. PMID 16329016
- [Result] Gondal G, Grotmol T, Hofstad B, Bretthauer M, Eide TJ, Hoff G. Lifestyle-related risk factors and chemoprevention for colorectal neoplasia: experience from the large-scale NORCCAP screening trial. Eur J Cancer Prev. 2005 Aug;14(4):373-9. doi: 10.1097/00008469-200508000-00010. PMID 16030428
- [Result] Skovlund E, Bretthauer M, Grotmol T, Larsen IK, Hoff G. Sensitivity of pain rating scales in an endoscopy trial. Clin J Pain. 2005 Jul-Aug;21(4):292-6. doi: 10.1097/01.ajp.0000110636.14355.3e. PMID 15951645
- [Result] Hoff G, Grotmol T, Thiis-Evensen E, Bretthauer M, Gondal G, Vatn MH. Testing for faecal calprotectin (PhiCal) in the Norwegian Colorectal Cancer Prevention trial on flexible sigmoidoscopy screening: comparison with an immunochemical test for occult blood (FlexSure OBT). Gut. 2004 Sep;53(9):1329-33. doi: 10.1136/gut.2004.039032. PMID 15306594
- [Result] Bretthauer M, Skovlund E, Grotmol T, Thiis-Evensen E, Gondal G, Huppertz-Hauss G, Efskind P, Hofstad B, Thorp Holmsen S, Eide TJ, Hoff G. Inter-endoscopist variation in polyp and neoplasia pick-up rates in flexible sigmoidoscopy screening for colorectal cancer. Scand J Gastroenterol. 2003 Dec;38(12):1268-74. doi: 10.1080/00365520310006513. PMID 14750648
- [Result] Bretthauer M, Hoff GS, Thiis-Evensen E, Huppertz-Hauss G, Skovlund E. Air and carbon dioxide volumes insufflated during colonoscopy. Gastrointest Endosc. 2003 Aug;58(2):203-6. doi: 10.1067/mge.2003.340. PMID 12872086
- [Result] Gondal G, Grotmol T, Hofstad B, Bretthauer M, Eide TJ, Hoff G. The Norwegian Colorectal Cancer Prevention (NORCCAP) screening study: baseline findings and implementations for clinical work-up in age groups 50-64 years. Scand J Gastroenterol. 2003 Jun;38(6):635-42. doi: 10.1080/00365520310003002. PMID 12825872
- [Result] Bretthauer M, Jorgensen A, Kristiansen BE, Hofstad B, Hoff G. Quality control in colorectal cancer screening: systematic microbiological investigation of endoscopes used in the NORCCAP (Norwegian Colorectal Cancer Prevention) trial. BMC Gastroenterol. 2003 Jun 13;3:15. doi: 10.1186/1471-230X-3-15. PMID 12803654
- [Result] Bretthauer M, Hoff G. The use of CO2 in colonoscopy. Gastrointest Endosc. 2003 Mar;57(3):436-7; author reply 437-8. doi: 10.1067/mge.2003.108. No abstract available. PMID 12612542
- [Result] Gondal G, Grotmol T, Hofstad B, Bretthauer M, Eide TJ, Hoff G. Grading of distal colorectal adenomas as predictors for proximal colonic neoplasia and choice of endoscope in population screening: experience from the Norwegian Colorectal Cancer Prevention study (NORCCAP). Gut. 2003 Mar;52(3):398-403. doi: 10.1136/gut.52.3.398. PMID 12584223
- [Result] Bretthauer M, Hoff G, Thiis-Evensen E, Grotmol T, Holmsen ST, Moritz V, Skovlund E. Carbon dioxide insufflation reduces discomfort due to flexible sigmoidoscopy in colorectal cancer screening. Scand J Gastroenterol. 2002 Sep;37(9):1103-7. doi: 10.1080/003655202320378329. PMID 12374237
- [Result] Bretthauer M, Hoff G, Thiis-Evensen E, Grotmol T, Larsen IK, Kjellevold O, Skovlund E. Use of a disposable sheath system for flexible sigmoidoscopy in decentralized colorectal cancer screening. Endoscopy. 2002 Oct;34(10):814-8. doi: 10.1055/s-2002-34273. PMID 12244504
- [Result] Larsen IK, Grotmol T, Bretthauer M, Gondal G, Huppertz-Hauss G, Hofstad B, Efskind P, Jorgensen A, Hoff G. Continuous evaluation of patient satisfaction in endoscopy centres. Scand J Gastroenterol. 2002 Jul;37(7):850-5. PMID 12190102
- [Result] Bretthauer M, Gondal G, Larsen K, Carlsen E, Eide TJ, Grotmol T, Skovlund E, Tveit KM, Vatn MH, Hoff G. Design, organization and management of a controlled population screening study for detection of colorectal neoplasia: attendance rates in the NORCCAP study (Norwegian Colorectal Cancer Prevention). Scand J Gastroenterol. 2002 May;37(5):568-73. doi: 10.1080/00365520252903125. PMID 12059059
- [Result] Bretthauer M, Thiis-Evensen E, Huppertz-Hauss G, Gisselsson L, Grotmol T, Skovlund E, Hoff G. NORCCAP (Norwegian colorectal cancer prevention): a randomised trial to assess the safety and efficacy of carbon dioxide versus air insufflation in colonoscopy. Gut. 2002 May;50(5):604-7. doi: 10.1136/gut.50.5.604. PMID 11950803
- [Derived] Jodal HC, Loberg M, Holme O, Adami HO, Bretthauer M, Emilsson L, Ransohoff DF, Hoff G, Kalager M. Mortality From Postscreening (Interval) Colorectal Cancers Is Comparable to That From Cancer in Unscreened Patients-A Randomized Sigmoidoscopy Trial. Gastroenterology. 2018 Dec;155(6):1787-1794.e3. doi: 10.1053/j.gastro.2018.08.035. Epub 2018 Aug 27. PMID 30165051
- [Derived] Holme O, Loberg M, Kalager M, Bretthauer M, Hernan MA, Aas E, Eide TJ, Skovlund E, Lekven J, Schneede J, Tveit KM, Vatn M, Ursin G, Hoff G; NORCCAP Study Groupdagger. Long-Term Effectiveness of Sigmoidoscopy Screening on Colorectal Cancer Incidence and Mortality in Women and Men: A Randomized Trial. Ann Intern Med. 2018 Jun 5;168(11):775-782. doi: 10.7326/M17-1441. Epub 2018 Apr 24. PMID 29710125
- [Derived] Berstad P, Botteri E, Larsen IK, Loberg M, Kalager M, Holme O, Bretthauer M, Hoff G. Lifestyle changes at middle age and mortality: a population-based prospective cohort study. J Epidemiol Community Health. 2017 Jan;71(1):59-66. doi: 10.1136/jech-2015-206760. Epub 2016 Jun 16. PMID 27312250
- [Derived] Swanson SA, Holme O, Loberg M, Kalager M, Bretthauer M, Hoff G, Aas E, Hernan MA. Bounding the per-protocol effect in randomized trials: an application to colorectal cancer screening. Trials. 2015 Nov 30;16:541. doi: 10.1186/s13063-015-1056-8. PMID 26620120
- [Derived] Riedel BM, Molloy AM, Meyer K, Fredriksen A, Ulvik A, Schneede J, Nexo E, Hoff G, Ueland PM. Transcobalamin polymorphism 67A->G, but not 776C->G, affects serum holotranscobalamin in a cohort of healthy middle-aged men and women. J Nutr. 2011 Oct;141(10):1784-90. doi: 10.3945/jn.111.141960. Epub 2011 Aug 24. PMID 21865561
- [Derived] Hoff G, Bretthauer M. Appointments timed in proximity to annual milestones and compliance with screening: randomised controlled trial. BMJ. 2008 Dec 17;337:a2794. doi: 10.1136/bmj.a2794. PMID 19091759
- See also: Website for the Norwegian Cancer Registry — http://www.kreftregisteret.no/en/